CLINICAL TRIAL: NCT06605690
Title: An Exploratory Clinical Study of Dalpiciclib an&Amp;#39;d Letrozole Combined With Anlotinib Neoadjuvant Therapy in Stage II-III Postmenopausal HR+/HER2- Early Breast Cancer
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Liu Shu (Other)
Responsible Party: Sponsor-Investigator, Liu Shu, Chief physician, The Affiliated Hospital Of Guizhou Medical University
Organization: The Affiliated Hospital Of Guizhou Medical University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Guizhou medical university
Record Dates: First submitted 2024-09-18; First posted 2024-09-20 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2024-09

CONDITIONS: Breast Cancer
Keywords: dalpiciclib;Anlotinib; Neoadjuvant Therapy HR+/HER2- Early Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — dalpiciclib; anlotinib

STUDY DESIGN:
Intervention Model Description: alpiciclib and Letrozole Combined With Anlotinib
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- experimental (Experimental): Dalpiciclib and Letrozole Combined With Anlotinib
  Interventions: Drug: Dalpiciclib and Letrozole Combined With Anlotinib

INTERVENTIONS:
Drug: Dalpiciclib and Letrozole Combined With Anlotinib — Dalpiciclib: 150mg orally, once daily, d1-d21, every 28 days as a cycle (3 weeks / 1 week off) Letrozole: 2.5mg orally once daily (continuous) Anlotinib: 12mg orally, once daily, d1-d14, every 21 days as a cycle (use 2 weeks/stop 1 week). One of the last cycles of the new auxiliary The combination of anlotinib is not included in the treatment regimen to ensure that the time interval between anlotinib withdrawal and surgery is more than 2-3 weeks.

SUMMARY:
This is a single-arm, open-label, exploratory clinical study

DETAILED DESCRIPTION:
This is a single-arm, open-label, exploratory clinical study initiated by the investigator to evaluate the objective response rate (ORR), efficacy, and safety of Dalpiciclib and letrozole combined with Anlotinib in the neoadjuvant treatment of stage Ⅱ-Ⅲ Postmenopausal HR+/HER2- breast cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Postmenopausal female patients, the definition of menopause:

(1) previous bilateral oophorectomy, or age ≥60 years; or(2) Age <60, natural postmenopausal status (defined as spontaneous cessation of regular menstruation for at least 12 consecutive months without other pathological or physiological causes), E2 and FSH in postmenopausal levels.

2. All patients had estrogen receptor (ER) positive (> 10%), HER2 receptor-negative invasive breast cancer regardless of PR expression level. Follow 2018 Asc-cap HER2 negative Interpretation guidelines. Immunohistochemical (IHC) score 0,1 + or 2+ and in situ hybridization (ISH) confirmed by pathology laboratory The test was negative (HER-2/CEP17 ratio < 2.0); 3. Patients with initial treatment of stage II-III whose tumor stage meets AJCC 8th edition standard; 4. No known severe hypersensitivity to chemical compounds or endocrine therapy similar to dalpiciclib or dalpiciclib excipients; Known against anlotinib or anlotinib Compounds with similar excipients had no severe hypersensitivity 5. ECOG 0-1; 6. The patient must have the ability to swallow oral drugs; 7. The level of organ function must meet the following requirements:

1. Bone marrow function ANC ≥ 1.5×109/L (no granulocyte stimulating factor was used within 14 days); PLT ≥ 100×109/L (no corrective therapy used within 7 days); Hb ≥ 100 g/L (no corrective therapy used within 7 days);
2. Liver and kidney function TBIL≤1.5×ULN;ALT and AST≤3×ULN (ALT and AST≤5×ULN in patients with liver metastasis);BUN and Cr≤1.5×ULN and creatinine clearance ≥50 mL/min (Cockcroft-Gault formula)
3. 12-lead electrocardiogram QT interval ≤480 ms; 8. Able to accept 2 puncture biopsies required by the protocol (puncture at the first diagnosis and puncture on the 15th day of medication) 9. Voluntarily participate in this study, sign informed consent, have good compliance and be willing to cooperate with follow-up.

Exclusion Criteria:

1. Previously received any form of anti-tumor therapy (chemotherapy, radiotherapy, molecular targeted therapy, endocrine therapy, etc.);
2. At the same time receive any anti-tumor treatment other than that prescribed in other protocols;
3. Bilateral breast cancer, inflammatory breast cancer or ocessive breast cancer;
4. Stage IV breast cancer;
5. Other malignant tumors have appeared in the past 5 years;
6. Severe heart, liver, kidney and other vital organ dysfunction;
7. Inability to swallow, chronic diarrhea, and intestinal obstruction, with multiple factors affecting drug use and absorption;
8. Known allergic history of the drug components of this protocol; Have a history of immunodeficiency, including HIV positive, HCV, active viral hepatitis B, or Have other acquired or congenital immunodeficiency diseases, or have a history of organ transplantation;
9. Pregnant and lactating women, women who are fertile and have a positive baseline pregnancy test or are unwilling to take effective treatment during the entire test period Female patients of reproductive age using contraceptives;
10. Concomitant diseases (including but not limited to uncontrollable drugs) that, in the judgment of the investigator, seriously endanger the patient's safety or interfere with the patient's completion of the study Severe hypertension, severe diabetes, active infection, etc.);
11. People with large risk of hemoptysis, such as patients with refractory hypertension; Blood system diseases such as idiopathic thrombocytopenic purpura, thrombocytopenia, etc.;Lung diseases such as active pulmonary tuberculosis and bronchiectasis; Patients with chronic liver disease such as cirrhosis, portal hypertension, etc., and other diseases that may present with massive hemoptysis disease;
12. Have a clear history of neurological or mental disorders, including epilepsy or dementia. The investigator did not consider the patient suitable for participation in any other condition of the study.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-10-31 (Estimated); Primary Completion 2025-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
ORR | 24 month
  Objective response rate